CLINICAL TRIAL: NCT04642911
Title: Longterm Follow-up of Subjects With Diabetes 2 Type Treatment With ex Vivo Gene Therapy Using Autologous Mesenchymal Stem Cell
Brief Title: Longterm Follow-up of Subjects With Diabetes 2 Type Treatment With ex Vivo Gene Therapy
Acronym: AUB001
Status: Active, not recruiting | Type: Observational
Sponsor: Ukraine Association of Biobank (Other)
Responsible Party: Sponsor
Other Study IDs: UAB00171120-1
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Diabete Type 2; Mesenchymal Stem Cell
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Long term follow up — Undergo long term follow up, including copy number measurement safety evaluations diseases specific product (Mesenchymal Stem Cell) in a Ukraine Association of Biobank bio-sponsored clinical trial who agree to participate in this study
  Other Names: LONG TERM; FOLLOW UP

SUMMARY:
This is a multicenter, long term safety and efficacy follow up study for with insulin dependent diabetes 2 type who have been treated with ex vivo gene therapy product in Ukraine Association of Biobank bio-sponsored clinical studies. After completing the parent clinical study (2 years),eligible subjects will be followed for an additional 8 years for total 10 years post-drugproduct infusion.

No investigation drug product will be administered in the study

ELIGIBILITY:
Inclusion Criteria:

* Treated with gene therapy of diabetes 2 type in a drug product (Mesenchymal Stem Cell) in a Ukraine Association of Biobank bio-sponsored clinical trial who agree to participate in this study
* Able to comply with study requirements
* Provision of written informed consent for this study by subjects or as applicable subject legal/parent guardian

Exclusion Criteria:

* There are no exclusion criteria for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject with diabetic 2 type who have treated with gene therapy in a drug product (Mesenchymal Stem Cell) in a Ukraine Association of Biobank bio-sponsored clinical trial who agree to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2030-10-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival of subject with diabetes 2 type with gene therapy drug product (Mesenchymal Stem Cell) in a Ukraine Association of Biobank bio-sponsored clinical trial who agree to participate in this study | 10 years post-drug product infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Bio-Stem Cell Rehabilitation, Kharkiv, Ukraine